CLINICAL TRIAL: NCT03055091
Title: Xylitol for the Prevention of Acute Otitis Media Episodes in Children 2-4: A Pragmatic RCT
Brief Title: Xylitol for the Prevention of Acute Otitis Media Episodes in Children
Acronym: POME-Xylitol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-300
Record Dates: First submitted 2017-02-03; First posted 2017-02-16 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Acute Otitis Media; URTI; Dental Caries in Children
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Intervention Model Description: This will be a pragmatic triple blind (participant and parents, practitioners and analyst will be blinded), two arm, superiority, placebo controlled randomized trial with 1:1 allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to the treatment arm or control arm and will receive the study product or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants in the treatment arm will receive a Xylitol syrup.
  Interventions: Other: Xylitol syrup
- Placebo (Placebo Comparator): Participants in the placebo arm will receive sorbitol syrup.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Xylitol syrup — Each dose will be 5 mL of 400 g/L and subjects will receive Three to 5 doses will be given each day.
  Arms: Treatment group
Other: Placebo — Each dose looks and tastes like the xylitol syrup but it is not microbial. Each dose will be 5 mL of 300 g/L of sorbitol. Three to 5 doses will be given each day.
  Other Names: Sorbitol syrup
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial of regular daily use of xylitol (or "birch sugar"), a natural sweetener that has antimicrobial properties, for the prevention of acute otitis media (AOM, primary outcome) as well as upper respiratory tract infections and dental caries (the two secondary outcomes) in preschool aged children. This trial will be conducted through the TARGet Kids! research network.

DETAILED DESCRIPTION:
This is an RCT of regular daily use of xylitol (or "birch sugar"), a natural sweetener that has antimicrobial properties, for the prevention of acute otitis media (AOM, primary outcome) as well as upper respiratory tract infections and dental caries (the two secondary outcomes) in preschool aged children. Clinical equipoise over the efficacy of xylitol in preventing AOM - a common and costly condition in early childhood - persists even after the completion of three RCTs by a single research group in Finland and one in the United States. Several clinical trials of xylitol for the prevention of dental caries and other studies have demonstrated that the intervention in this trial (3-5 doses of xylitol per day) is safe, well tolerated and feasible for the study period. This trial will be conducted through the TARGet Kids! research network which is undertaking several CIHR funded RCTs and will leverage existing CIHR funded infrastructure and important collaborations. The nominated principal applicant's salary is supported by a CIHR RCT training grant to develop this RCT under the mentorship of a co-principal applicant who is an experienced trialist. This trial has the potential to transform the management of three common conditions during early childhood from treatment to prevention using a currently underutilized antimicrobial substance.

ELIGIBILITY:
Inclusion Criteria:

* Children already enrolled in the TARGet Kids! Network, age 2 - 4 years at start of intervention, parents or care provider able to give consent, able to understand the information in English.

Exclusion Criteria:

* craniofacial malformations, structural middle ear abnormalities, sibling or any other child living at the same address already enrolled in the trial, insertion of ventilation tubes prior to study period, current use of a xylitol product or reported xylitol sensitivity.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 472 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
acute otitis media episodes | 6 months
  Total number of physician diagnosed acute otitis media episodes

SECONDARY OUTCOMES:
upper respiratory tract infection episodes | 6 months
  Total number of parent or caregiver reported upper respiratory tract infection episodes
dental caries | 6 months
  absence of dental caries by parent report

OTHER OUTCOMES:
costs to parents including costs associated with attending medical appointments related to acute otitis media and lost productivity | 6 months
  the costs of attending medical appointment will include the cost of transportation and the mode of transportation will be asked during a monthly call

CONTACTS AND LOCATIONS:
Overall Officials: Nav Persaud, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persaud N, Azarpazhooh A, Keown-Stoneman C, Birken CS, Isaranuwatchai W, Maguire JL, Mamdani M, Allen C, Mason D, Kowal C, Jaleel M, Bazeghi F, Thorpe KE, Laupacis A, Parkin PC. Xylitol for the prevention of acute otitis media episodes in children aged 1-5 years: a randomised controlled trial. Arch Dis Child. 2024 Jan 22;109(2):121-124. doi: 10.1136/archdischild-2023-325565. PMID 37890960
- [Derived] Persaud N, Laupacis A, Azarpazhooh A, Birken C, Hoch JS, Isaranuwatchai W, Maguire JL, Mamdani MM, Thorpe K, Allen C, Mason D, Kowal C, Bazeghi F, Parkin P; TARGet Kids! Collaboration. Xylitol for the prevention of acute otitis media episodes in children aged 2-4 years: protocol for a pragmatic randomised controlled trial. BMJ Open. 2018 Aug 5;8(8):e020941. doi: 10.1136/bmjopen-2017-020941. PMID 30082349
- See also: The Applied Research Group — http://TARGETKIDS.CA